CLINICAL TRIAL: NCT01501526
Title: Unusual Clinical Findings of Herpes Esophagitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DMR100-IRB-190
Record Dates: First submitted 2011-12-25; First posted 2011-12-29 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Herpes Esophagitis; Vocal Fold Palsy
Keywords: herpes esophagitis; dysphagia; vocal fold palsy; immunocompetent; husky voice
MeSH Terms: conditions — Vocal Cord Paralysis; Deglutition Disorders; Dysphonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Herpes esophagitis presents a clinical diagnostic challenge. The investigators report the first case of herpes esophagitis presenting as vocal fold palsy in an immunocompetent host. The investigators case highlights the importance of performing a detailed laryngoscopic examination in any patient with prolonged husky voice.

ELIGIBILITY:
Inclusion Criteria:

* Patient of Herpes esophagitis with vocal palsy presentation

Exclusion Criteria:

* Patient of Herpes esophagitis without vocal palsy presentation

Ages: 50 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2011-10; Study Completion 2012-03 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan, Taiwan